CLINICAL TRIAL: NCT06539923
Title: Sarcopenic Index and Related Factors in Patients With Type 2 Diabetes Applying to Tertiary Health Care Services
Brief Title: Sarcopenic Index and Related Factors in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, Ayse N Erbakan, Principal İnvestigator, Goztepe Prof Dr Suleyman Yalcın City Hospital
Other Study IDs: SI in T2DM
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes; Sarcopenia
Keywords: type 2 diabetes; sarcopenic index; Cystatin C
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- T2DM patients: patients with definite type 2 diabetes diagnosis
  Interventions: Other: retrieving data

INTERVENTIONS:
Other: retrieving data — Data will be retrieved retrospectively

SUMMARY:
Sarcopenia, characterized by a progressive loss of skeletal muscle mass and function, is particularly common in individuals with T2DM and is often associated with insulin resistance, chronic inflammation and oxidative stress. The Sarcopenia Index (SI), calculated as serum creatinine divided by serum cystatin C, is a practical tool for assessing sarcopenia and is used in many clinical settings. In this study, we aimed to investigate the relationship between sarcopenic index and variables such as age, diabetes duration, diabetes control and complication-related parameters such as NT-proBNP and Fib4 score in patients with type 2 diabetes.

DETAILED DESCRIPTION:
This study was planned retrospectively. Between September 01, 2023 and March 31, 2024, the records of patients who presented to the Diabetes Outpatient Clinic of Goztepe Prof. Dr. Suleyman Yalcin City Hospital for Internal Medicine and whose routine biochemical tests (including NT-proBNP and cystatin C) were found in the system will be retrospectively reviewed. Both male and female patients with a definite diagnosis of type 2 diabetes were included in the study. Inclusion criteria included: age 40 years or older, age 85 years or younger, no acute infection, no steroid use, no acute changes in creatinine or cystatin C levels, no recent surgery, no limb loss. Demographic data included age, gender, duration of diabetes, medications and concomitant diseases. The Fib 4 score was calculated using the patients' routine biochemical and hematologic results. The sarcopenia index was calculated from the serum creatinine/cystatin C values. A cut-off value of 0.90 is normally used for the diagnosis of sarcopenia in people without diabetes, but there is no cut-off value for patients with diabetes. Therefore, in addition to the correlation, the SI value was divided into 3 groups and the patients in the lowest and highest groups were compared with each other.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes diagnosis
* with complete biochemical data on record

Exclusion Criteria:

* acute infection,
* steroid use,
* acute changes in creatinine or cystatin C levels,
* recent surgery,
* limb loss.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were diagnosed with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 839 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Age | baseline
  relationship between sarcopenic index and age
diabetes duration | baseline
  relationship between sarcopenic index and diabetes duration
Glycemic control | baseline
  relationship between sarcopenic index and glycemic control using HbA1c levels
NT-proBNP | baseline
  relationship between sarcopenic index and NT-proBNP (NT terminal pro-brain natriuretic peptide-use for assessing heart failure) levels
FIB4 score | baseline
  relationship between sarcopenic index and Fib4 score ( reflecting hepatic fibrosis risk)

CONTACTS AND LOCATIONS:
Overall Officials: Ayse N Erbakan, MD, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- SB Istanbul Goztepe Prof Dr Suleyman Yalcin City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No